CLINICAL TRIAL: NCT04008524
Title: A Clinical Study of CAR-T Cells in the Treatment of Relapsed and Refractory Hematological Malignancies
Status: Available | Type: Expanded Access
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: QT2019006
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-02

CONDITIONS: Relapsed and Refractory Hematological Malignancies
Keywords: Relapsed; Refractory; Hematological malignancy; CAR-T cells
MeSH Terms: conditions — Recurrence; Hematologic Neoplasms | interventions — Immunotherapy, Adoptive

INTERVENTIONS:
Biological: CAR-T cells — Chimeric Antigen Receptor-T cells

SUMMARY:
This project is intended to provide CAR-T cell therapy products for patients with severely life-threatening relapsed and refractory hematological malignancies. These patients have been previously treated sufficiently, currently have no other treatment methods available, and do not meet the inclusion criteria of other clinical trial projects in the process of subject recruitment or meet their exclusion criteria. This project is designed to meet the urgent clinical needs of individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from a hematological malignancy that is severely life-threatening or seriously affects the patient's quality of life and has no effective treatment available, who not meet the inclusion/exclusion criteria for other clinical trials in the process of subject recruitment, or who are unable to obtain other study drugs or participate in clinical studies/trials for some reason (regional or time restriction, etc., or the recruitment of subjects for clinical studies/trials has ended but the drug has not yet been approved for marketing in China);
* Patients who are definitely diagnosed with the corresponding target-positive relapsed and refractory hematological malignancies, including but not limited to the following circumstances:

  * Patients who do not meet the inclusion/exclusion criteria for existing clinical trials, such as age <18 years, ECOG >1, extramedullary recurrence, persistent or repeatedly positive for minimal residual disease;
  * Patients who have relapsed after remission following CAR-T cell therapy, and are expected as judged by the investigator to benefit more from re-use of the same cell or sequential use of other CAR-T cells compared with the risk;
  * The quantity of CAR-T cells produced does not meet the release criteria of production quality inspection, but is >0.1× 106/kg CAR positive T cells, and the investigator judges that the expected benefit of cell infusion is greater than the risk;
  * The disease progresses rapidly after cell collection and before infusion, and the investigator judges that the expected benefit of cell infusion is greater than the risk;
  * Patients who have relapsed after autologous/heterogeneous hematopoietic stem cell transplantation (including those positive for minimal residual disease);
  * Other circumstances where the investigator judges that the expected benefit of cell infusion is greater than the risk.
* Patients with appropriate bone marrow reserve: such as lymphocyte count >0.3×109/L;
* Patients with proper heart, lung, liver, kidney and coagulation functions;
* The selected patients or their legal representatives voluntarily sign the informed consent form.

Exclusion Criteria:

* Patients who are positive for any of HIV antibody, TP antibody, HBsAg and HCV antibody.
* Patients with a history of epilepsy or other central nervous system diseases.
* Patients with evidence of currently uncontrollable serious active infections (e.g., sepsis, bacteremia, fungemia, viremia, etc.).
* Patients with other conditions making the patients unsuitable for receiving cell therapy as judged by the investigator.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, China